CLINICAL TRIAL: NCT01355172
Title: Clinical Study Protocol Immunogenicity and Safety of a Trivalent Inactivated Influenza Vaccine, Formulation 2010-2011， in Infants Aged Between 6-12months Old
Brief Title: Immunogenicity and Safety of AdimFlu-S, Formulation 2010-2011, in Infants Aged Between 6-12months Old
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Adimmune Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: FLU10T11C
Record Dates: First submitted 2011-05-15; First posted 2011-05-18 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Influenza
Keywords: Influenza; Vaccine; Immunogenicity
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: AdimFlu-S — 0.25mL per injection 2 injections at 4 weeks apart

SUMMARY:
The purpose of this study is to evaluate the antibody response to each of the three influenza vaccine strains included in the seasonal flu vaccine(AdimFlu-S), as measured by hemagglutination inhibition (HAI) at 4 weeks after two doses of study vaccine, 4 weeks apart, in infants between 6 and 12 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Boys or girls and aged >= 6 months old to <= 12 months old on the day of first vaccination;
* Subject's parent(s) or legal guardian(s) must be willing to comply with planned study procedures and be available for all study visits;
* Subject must be in good physical health on the basis of medical history, physical examination;
* Subject's parent(s) or legal guardian(s) must read and signed the study-specific informed consent prior to initiation of any study procedure.

Exclusion Criteria:

* Subjects had received influenza vaccine;
* History of hypersensitivity to eggs or egg protein or similar pharmacological effects to study medication;
* Personal or family history of Guillain- Barre' Syndrome;
* An acute febrile illness within 1 week prior to vaccination;
* Current upper respiratory illness (URI), including the common cold or nasal congestion within 72 hours;
* Subjects with influenza-like illness as defined by the presence of fever (temperature >= 38'C) and at least two of the following four symptoms: headache, muscle/joint aches and pains (e.g. myalgia/arthralgia), sore throat and cough;Treatment with an investigational drug or device, or participation in a clinical study, within 3 months before consent;
* Immunodeficiency, immunosuppressive or significant chronic illness not suitable for inactivated influenza vaccination;
* History of wheezing or bronchodilator use within 3 months prior to study vaccine;
* Receipt of live virus vaccine within 1 month prior to study vaccine or expected receipt vaccination before the last blood sampling for immunogenicity evaluation;
* Receipt of any inactivated vaccine within 2 weeks prior to study vaccination or expected receipt vaccination before the last blood sampling for immunogenicity evaluation;
* Receipt of any blood products, including immunoglobulin in the prior 3 months;
* Underlying condition in the investigators' opinion may interfere with evaluation of the vaccine.

Ages: 6 Months to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2010-11; Primary Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
HA antibody titers will be determined using the WHO HAI reference technique. | Serum samples will be obtained prior to vaccination (baseline), and 4 weeks after each vaccination.

SECONDARY OUTCOMES:
The secondary objective is to evaluate the safety and tolerability profiles including the presence or absence of the pre-specified reactogenicity events and other serious/non-serious adverse events of the AdimFlu-S manufactured by Adimmune Corporation. | (4 weeks after two doses of study vaccine, 4 weeks apart), Physical examination will be performed at each visit. Reactogenicity will be recorded for 7 days after each vaccination.
  Safety data will consist of reactogenicity, serious and non-serious adverse events. Reactogenicity events are pre-specified adverse events systematically recorded for 7 days after each vaccination.
  The events included fever (≥38.0°C), runny nose or nasal congestion, cough, sore throat, muscle aches, headache, vomiting, nausea and malaise. Furthermore, the local (injection site) reactions were also evaluated, including soreness/pain, swelling, redness, ecchymosis and limitation of arm motion.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medicine University Hospital, Taichung, Taiwan